CLINICAL TRIAL: NCT01110109
Title: EVAC Use in the OR: A Randomized Clinical Study to Evaluate the Content of Fluid Extracted From the Endotracheal Tube Cuff Using Intermittent and Continuous Suctioning During Surgery
Brief Title: Removing Fluid Above Breathing Tubes in the Operating Room
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Jonathan Bissett/Clinical Research Associate II, Covidien
Other Study IDs: COV-MO-PO-A111
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Adult; Surgery; Endotracheal Tube; Ventilator; Pneumonia; Suctioning
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Suction secretions
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Continuous Suctioning: Anesthesia staff will suction secretions continuously at 20 mmHg with a safety stop of 5 seconds every 30 minutes.
- Intermittent Suctioning: Anesthesia staff will suction secretions intermittently using an intermittent suction regulator. The regulator will be set to suction at 100-150 mmHg. The regulator has a preset cycle of intermittent suctioning for 15 seconds with an 8 second pause.

SUMMARY:
In this study, subjects meeting criteria will be enrolled and randomized to one of two different suctioning schemes, either continuous or intermittent. Accumulated secretions will be collected above the cuff on the breathing tube by one of the two methods depending on which group the subject is randomized into. Secretions will continue to be collected at predetermined periods of time for the duration of surgery in order to characterize the pH and volume as well as the micro-organism content.

DETAILED DESCRIPTION:
The development of pneumonia and other infections from intubation in the intraoperative setting has not been well-studied. An understanding of the content of the fluid that accumulates above the cuff in this setting will further strengthen the relationship between intubation and infection. The purpose of this study is to characterize the content of fluid extracted from the endotracheal tube cuff during surgery. This study will also evaluate the content of the fluid across various intervals of suctioning.

Suctioning Schemes -

* Continuous Suctioning Anesthesia staff will suction secretions continuously at 20 mmHg with a safety stop of 5 seconds every 30 minutes. Staff will be responsible for monitoring the interval between each safety stop.
* Intermittent Suctioning Anesthesia staff will suction secretions intermittently using an intermittent suction regulator. The regulator will be set to suction at 100-150 mmHg. The regulator has a preset cycle of intermittent suctioning for 15 seconds with an 8 second pause.

This is a prospective randomized clinical study of 48 subjects at a single site in the United States. Those placing the tube and performing the suctioning schemes will be experienced study staff and have met all training requirements to ensure consistency. Subjects will be patients undergoing surgery requiring intubation using the TaperGuard Evac Endotracheal Tube for a minimum of two hours, but no longer than twelve hours. They must also be 18 years of age or older, able to provide consent and have no presence of tracheostomy. Pregnant subjects will also be excluded.

Suctioning will begin as soon as the tube is in place and will continue until extubation or until the patient is moved from the operating room, whichever comes earlier. Secretions will be collected in a Lukens Trap. Anesthesia staff will collect the accumulated secretions every 30 minutes for the duration of the surgery, and secretions will be processed according to the instructions provided in the sample collection kit.

To address the first objective of the study, the first and last sample obtained from each subject will be analyzed individually for pH, volume, and microorganisms; all other samples will be evaluated for volume. The amount of colony forming units (CFUs) will be determined semi-quantitatively across all organisms, and presented separately for individual genera and species. The samples will be characterized with descriptive statistics including frequencies, percentages, means, medians, standard deviations, and 95% CIs. To address the second objective of the study, comparisons of pH, volume, microorganisms, and CFUs by suctioning scheme and patient-level characteristics will be conducted using chi-squared tests of independence and analysis of variance (ANOVA). Graphical methods will be developed to aid interpretation, both as a function of time and cumulatively over time.

ELIGIBILITY:
Inclusion Criteria:

* Surgery to be performed with expected time between tracheal intubation and extubation of at least two hours, but no longer than 12 hours
* Intubation planned with TaperGuard EVAC Endotracheal Tube
* Age of 18 or older
* Ability to provide informed consent

Exclusion Criteria:

* Presence of tracheostomy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing surgery requiring intubation using the TaperGuard EVAC Endotracehal Tube
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis A Rosinia, M.D., Principal Investigator — Tulane University Hospital
Locations (1):
- Tulane University Hospital, New Orleans, Louisiana, United States